CLINICAL TRIAL: NCT00799136
Title: Feasibility Study of CO-administering Combination Antiretroviral Therapy (cART) and R-EPOCH Chemotherapy for the Management of Acquired Immunodeficiency Syndrome (AIDS)-Related Lymphoma
Brief Title: A Feasibility Study of Co-administering Combination Antiretroviral Therapy (cART) and R-EPOCH Chemotherapy for the Management of ARL
Acronym: CATCH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCOG-2007-CATCH; CIHR FRN 79390
Record Dates: First submitted 2008-11-26; First posted 2008-11-27 (Estimated); Last update posted 2013-09-12 (Estimated); Status verified 2013-09

CONDITIONS: Lymphoma, AIDS Related; HIV Infections
Keywords: Lymphoma Large B Cell Diffuse; Acquired Immunodeficiency
MeSH Terms: conditions — Lymphoma, AIDS-Related; HIV Infections; Dendritic Cell Sarcoma, Interdigitating | interventions — Rituximab; Etoposide; Doxorubicin; Vincristine; Cyclophosphamide; Prednisone; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- One (Other): Rituxan with EPOCH and Antiretrovirals
  Interventions: Drug: R-EPOCH and cART

INTERVENTIONS:
Drug: R-EPOCH and cART — This is a prospective, single-arm, multi-centre, phase II trial of immuno-chemotherapy (rituximab and EPOCH) with mandatory combination antiretroviral therapy for initial treatment of AIDS-related lymphoma.
  Other Names: Rituxan; Vepesid; Adriamycin; Vincristine; Cytoxan; Prednisone; Truvada; Sustiva

SUMMARY:
No standard regimen currently exists for the treatment of AIDS-related lymphoma. Based on the encouraging NCI results with DA-EPOCH, the US AIDS Malignancy Consortium is currently administering a phase II randomized protocol comparing EPOCH with sequential versus concurrent rituximab (AMC protocol 034). In this AMC trial, the decision to co-administer cART is left to the discretion of the treating physician and the patient. While the AMC phase II study may establish an acceptable chemotherapy regimen suitable for further study in a phase III randomized trial, the results will not address adherence, pharmacokinetic interactions or the role of cART in AIDS-related lymphoma. The contribution of cART to the anti-lymphoma efficacy of any regimen needs to be formally studied. Our proposed trial to demonstrate the feasibility of co-administering cART with chemotherapy would justify the use of combined therapy in future AMC/International phase III protocols.

DETAILED DESCRIPTION:
Study Design & Duration This is a prospective, single-arm, multi-centre, phase II trial of immuno-chemotherapy (rituximab and EPOCH) with mandatory combination antiretroviral therapy for initial treatment of AIDS-related lymphoma. Patients diagnosed with previously-untreated AIDS-related diffuse large B-cell lymphoma will be eligible for this trial. Patients are eligible regardless of whether they have previously been treated with or are naïve to antiretroviral therapy. The total sample size of 18 patients is required to determine the feasibility of co-administering cART and chemotherapy as measured by adequate adherence to the antiretroviral regimen.

Patients will receive EPOCH and rituximab chemotherapy for 6 cycles each given every 21 days. Day 1 of each cycle will consist of an infusion of rituximab followed by the initiation of a 96-hour continuous infusion of etoposide, doxorubicin, and vincristine and oral prednisone. Cyclophosphamide will be administered on Day 5 with initial dose based on initial CD4+ cell count to minimize hematologic toxicity.

Combination antiretroviral therapy will be administered to all patients enrolled in the trial. Patients already responding to their current cART regimen will continue with the same therapy. Otherwise, patients can be initiated on a preferred regimen of tenofovir (TDF), emtricitabine (FTC), and efavirenz (EFV) according to the US Department of Health and Human Services (DHHS) guidelines. Patients initiated on the preferred regimen of TDF/FTC/EFV will start the antiretroviral treatments on Day 7 of the trial, after the first cycle of R-EPOCH is administered. Treatment will subsequently be continued for the duration of the trial and thereafter, according to the discretion of the treating physician.

The primary endpoint for this feasibility study will be medication adherence to cART treatment. "Acceptable adherence" will be defined as the proportion of patients able to complete >90% of all prescribed cART doses during the course of chemotherapy as measured by pill counts. As previously reported, study participants will be asked to bring their pill bottles to clinic prior to each chemotherapy cycle (every three weeks) so that remaining pills can be counted by the participating study nurse/pharmacist. The number of missed doses will be computed from the difference between the actual and expected number of pills remaining in the bottle. Secondary outcomes include the toxicity of the combination therapy, as measured by adverse events graded according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0. CD4+ cell counts and HIV-1 mRNA viral loads will be obtained on all patients at baseline, following recovery from cycles 3 and 6, and every three months thereafter for two years. Secondary outcomes will also include complete and partial lymphoma response rate, progression-free survival, and overall survival, all defined by International Working Group criteria. The pharmacokinetics of etoposide, vincristine and doxorubicin will be studied in the patients initiating the preferred antiretrovirals TDF/3TC/EFV on Day 7 of the protocol (after completion of the first cycle of R-EPOCH). Thus the analysis of PK interactions will be on this subgroup of patients receiving a uniform treatment strategy. Pharmacokinetics will be assessed with the first cycle (when chemotherapy is given alone) and subsequent cycle of R-EPOCH (when chemotherapy is given with cART).

Study administration and data collection will occur under the auspices of the Ontario Clinical Oncology Group (OCOG). OCOG operates from within the Clinical Trials Methodology Group at the Henderson Research Centre in Hamilton and is co-directed by oncologists at the Juravinski Cancer Centre and Toronto Sunnybrook Cancer Centres. OCOG has a well-established research environment to guide the administration of this trial across four unique clinical sites across Canada. The clinical sites for the study include Toronto Sunnybrook Regional Cancer Centre (TSRCC), Princess Margaret Hospital (PMH), St. Michael's Hospital (SMH), and at the St. Paul's Hospital (SPH) in Vancouver. Each clinical site is expected to enroll 1-4 patients per year. An overall accrual rate of 8-10 patients per year is expected. Therefore, it will be possible to register 18 patients within 2 years of study initiation. For the individual patient, the chemotherapy treatment duration is 18 weeks. Following this phase of therapy (18 weeks), individual patients will be followed every 3 months for an additional 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. HIV seropositivity
2. Biopsy diagnosis of a CD20+ diffuse large B-cell lymphoma or variants (including mediastinal (thymic) large B-cell lymphoma and plasmablastic lymphoma), atypical Burkit/Burkitt-like lymphoma, or Burkitt lymphoma diagnosed according to the World Health Organization (WHO) classification
3. Age 18 years or older

Exclusion Criteria

1. Performance status ≥3 according to ECOG (Zubrod) scale (see Appendix I)
2. Known primary central nervous system lymphoma or parenchymal brain involvement with lymphoma
3. Non-measurable disease by physical examination or radiographic evaluation
4. Absolute CD4+ cell count <50 cells/mm3 within 3 months prior to trial initiation
5. Inadequate hepatic function (total bilirubin ≥35 µmol/L, alkaline phosphatase ≥2 xUL normal, AST/ALT ≥2 xUL normal) unless directly attributable to lymphoma or known Hepatitis B or C co-infection.
6. Inadequate renal function (serum creatinine ≥125µmol/L) unless directly attributable to lymphoma
7. Inadequate haematological function (haemoglobin ≤85 g/L, absolute neutrophil count ≤1000 cells/mm3, platelet count ≤75,000 cells/mm3) unless directly attributable to lymphoma or autoimmune thrombocytopenia.
8. Evidence of left ventricular (LV) dysfunction (ejection fraction ≤ 50%) in patients over the age of 60 or in patients with a prior history of hypertension, congestive heart failure, peripheral vascular disease, cerebrovascular disease, coronary artery disease, or cardiac arrhythmia
9. Pregnant or lactating women who intend to breast-feed during the trial period
10. Men of reproductive potential and women of childbearing potential who are not using or not willing to use effective contraception
11. Known intolerance to the prescribed chemotherapy or antiretroviral drugs
12. Life-expectancy ≤ 3 months
13. Geographically inaccessible for follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-02; Primary Completion 2012-12 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
The primary outcome for this feasibility study will be medication adherence. Acceptable adherence, defined as compliance to ≥90% of all prescribed doses of cART during the course of chemotherapy, will be measured by pill counting and patient self-report | 4 -6 weeks after 6 cycles of R-EPOCH

SECONDARY OUTCOMES:
Toxicity Lymphoma response Rate Progression -free Survival and Overall Survival Pharmacokinetics | 2 years post completion

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Cheung, Dr. ., Principal Investigator — Odette Cancer Centre
Locations (2):
- Canada (2):
  - Odette Cancer Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario